CLINICAL TRIAL: NCT04747275
Title: Use of Liquid Stable Levothyroxine in Trisomy 21 Pediatric Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Transitioned to multi site study with sponsor
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Matthew Feldt, Physician, DO, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY00001385
Record Dates: First submitted 2021-02-03; First posted 2021-02-10 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Hypothyroidism; Trisomy 21
Keywords: Tolerability; Adherence
MeSH Terms: conditions — Hypothyroidism; Down Syndrome | interventions — Thyroxine

STUDY DESIGN:
Intervention Model Description: Phase 4, single-center, pilot, randomized, open-label, cross-over study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liquid Stable Levothyroxine (l-T4) TirosintSOL first, then Oral Tablet Levothyroxine (L-T4) (Other): Participants start on Liquid Tirosint®-SOL for 8 weeks using continued same daily dose of LT4. Dose adjustments are allowed as needed, based on laboratory results and clinical response. Then Participants will crossover to conventional therapy of LT4 tablets for 8 weeks. Participants total participation will be 16 weeks total.
  Interventions: Drug: Liquid stable levothyroxine (L-T4) Tirosint-SOL; Drug: Oral tablet levothyroxine (L-T4)
- Oral Tablet Levothyroxine (L-T4) first, then Liquid Stable Levothyroxine (L-T4) Tirosint-SOL (Other): Participants continue conventional therapy of LT4 tablets for 8 weeks at current dose, after 8 weeks will crossover to receive Liquid Stable Levothyroxine (L-T4) Tirosint-SOL for 8 weeks. Participants total participation will be 16 weeks total.
  Interventions: Drug: Liquid stable levothyroxine (L-T4) Tirosint-SOL; Drug: Oral tablet levothyroxine (L-T4)

INTERVENTIONS:
Drug: Liquid stable levothyroxine (L-T4) Tirosint-SOL — Investigation of tolerability, palatability, and adherence of liquid levothyroxine (L-T4) for 8 weeks.
Drug: Oral tablet levothyroxine (L-T4) — Investigation of tolerability, palatability, and adherence of maintained oral tablet levothyroxine (L-T4) for 8 weeks

SUMMARY:
Children with levothyroxine (T21) have developmental delay and other functional gastrointestinal (GI) issues that may negatively affect L-T4 tolerability and absorption. For an age group unable to swallow tablets whole by mouth, tablets must be crushed and suspended in water, breast milk or formula for administration in order to treat children with hypothyroidism. For this age group, ease of administration may have a significant impact on compliance and ability to remain euthyroid. We propose that Tirosint-SOL® will be more favorably received due to ease of administration, improved tolerability and palatability, therefore leading to improved adherence when compared to L-T4 tablets.

DETAILED DESCRIPTION:
Hypothyroidism is a common medical disorder in children with Trisomy 21 (T21). Treatment with oral tablet levothyroxine (L-T4) is primarily used to treat this condition. However, children with T21 have developmental delay and other functional gastrointestinal (GI) issues that may negatively affect L-T4 tolerability and absorption. For an age group unable to swallow tablets whole by mouth, tablets must be crushed and suspended in water, breast milk or formula for administration in order to treat children with hypothyroidism. For this age group, ease of administration may have a significant impact on compliance and ability to remain euthyroid. Until recently, there was no liquid preparation of L-T4 in the United States for use in children. Tirosint-SOL® (liquid stable L-T4) is now FDA-approved for use in children. The Investigator proposes that Tirosint-SOL® will be more favorably received due to ease of administration, improved tolerability and palatability, therefore leading to improved adherence when compared to L-T4 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Trisomy 21 children age 2 months to less than 5 years of age
* Prior confirmed diagnosis of congenital or acquired hypothyroidism

Exclusion Criteria:

* Gestational age ≤ 35 weeks, concomitant anticonvulsant medications, history of nonadherence with medication or medical visit schedule
* Subjects must be able to take oral medication, no G-tube or parental fed subjects

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liquid Stable Levothyroxine (l-T4) TirosintSOL First, Then Oral Tablet Levothyroxine (L-T4) | Oral Tablet Levothyroxine (L-T4) First, Then Liquid Stable Levothyroxine (L-T4) Tirosint-SOL
Started | 2 | 4
Completed | 2 | 3
Not Completed | 0 | 1
Not completed — Study terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: 6 subjects were enrolled and completed the study, however, due to concerns with data collection and integrity, we elected to not use those subjects data moving forward. No further subjects were recruited prior to the study closing
Groups:
- Total: Total of all reporting groups
Arm/Group | Liquid Stable Levothyroxine (l-T4) TirosintSOL First, Then Oral Tablet Levothyroxine (L-T4) | Oral Tablet Levothyroxine (L-T4) First, Then Liquid Stable Levothyroxine (L-T4) Tirosint-SOL | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 4 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Tolerability as Assessed by the CareCAT Tool
Description: Utilize medication tolerability questionnaire, Care Children's Acceptance Tool (CAT), to understand parental perceptions of liquid stable L-T4.
Time Frame: 4 months
Population: 6 subjects were enrolled and 5 completed the study, however, due to concerns with data collection and integrity, the overseeing Institutional Review Board determined that results for these subjects should not be analyzed. No further subjects were recruited prior to the study closing.
Groups:
- Treatment: Participants started on Tirosint®-SOL using continued same daily dose of LT4. Dose adjustments are allowed as needed, based on laboratory results and clinical response. Participants will be treated for 16 weeks total.
- Control: Participants continue conventional therapy of LT4 tablets for 8 weeks at current dose, after 8 weeks will crossover to receive the treatment arm (Tirosint-SOL) for 8 weeks. Participants will be treated for 16 weeks total.
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Adherence to Taking Study Medication
Description: Evaluate differences in compliance with liquid stable L-T4 compared to L-T4 tablet. Evaluated in percentage of days compliant.
Time Frame: 4 months
Population: as for outcome 1
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 112 Days, Duration of Study.
Arm/Group | Liquid Stable Levothyroxine (l-T4) TirosintSOL First, Then Oral Tablet Levothyroxine (L-T4) | Oral Tablet Levothyroxine (L-T4) First, Then Liquid Stable Levothyroxine (L-T4) Tirosint-SOL
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 0/2 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT04747275/Prot_002.pdf
  • Informed Consent Form (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04747275/ICF_001.pdf